CLINICAL TRIAL: NCT00610454
Title: Trial Evaluating the Safety and Tolerability of Levetiracetam Intravenous 15-minute Infusion, Administered in b.i.d. Regimen as an Adjunctive Antiepileptic Treatment in Subjects From 16 to 65 Years Suffering From Partial Onset Seizures
Brief Title: Safety and Tolerability of Levetiracetam Intravenous 15 Minute Infusion in Subjects Suffering From Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01166
Record Dates: First submitted 2008-01-18; First posted 2008-02-08 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
Subjects receiving LEV as adjunctive therapy to 1 or 2 other AEDs for partial onset seizures and subjects who are temporarily unable to take oral LEV, may require alternative routes of administration. The purpose of this trial was to evaluate the safety and tolerability of 1000 to 3000 mg/day LEV administered as a 15-min IV infusion b.i.d. after switching from the same oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* in- or out-subjects suffering from partial onset seizures according to the ILAE classification of Epileptic Seizures;
* intake of levetiracetam as an adjunctive antiepileptic oral treatment in addition to one or two antiepileptic drugs (AED).

Exclusion Criteria:

* Had problems of venous accessibility;
* showed safety issues related to the administration of one of the concomitant AEDs requiring medical intervention;
* clinically significant ECG/lab abnormalities;
* administered vigabatrine;
* administered felbamate for less than 18 months;
* had contraindication to any component of the study medication treatment as IV formulation or known allergic reaction to or intolerance of pyrrolidone derivatives.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-06; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of levetiracetam after switching from oral formulation to 15-minute IV infusion during repeated dosing (4 days b.i.d.) | Adverse events after each infusion

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- [Background] Baulac M, Brodie MJ, Elger CE, Krakow K, Stockis A, Meyvisch P, Falter U. Levetiracetam intravenous infusion as an alternative to oral dosing in patients with partial-onset seizures. Epilepsia. 2007 Mar;48(3):589-92. doi: 10.1111/j.1528-1167.2006.00959.x. Epub 2007 Feb 22. PMID 17326794